CLINICAL TRIAL: NCT01627015
Title: Safety, Acceptance and Metabolic Effects in Infants Receiving a Novel Low Glycaemic Index follow-on Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Principal Investigator, Koletzko - Office, Prof. Berthold Koletzko, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 114-12
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Infant Nutrition
Keywords: Fully formula fed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified infant follow-on formula (Experimental): Infants are fed a modified infant follow-on formula (modified carbohydrate composition) for 4 weeks, according to protocol
  Interventions: Other: Modified infant follow-on formula
- Standard infant follow-on formula (Active Comparator): Infants are fed a commercial follow-on formula for 4 weeks, according to protocol
  Interventions: Other: Standard infant follow-on formula

INTERVENTIONS:
Other: Modified infant follow-on formula — The modified infant follow-on formula has a different carbohydrate pattern than the standard formula
  Arms: Modified infant follow-on formula
Other: Standard infant follow-on formula — Infants are fed a commercial follow-on formula
  Arms: Standard infant follow-on formula

SUMMARY:
In this study, the safety, acceptance and metabolic effects in infants receiving a novel low glycaemic index follow-on formula will be investigated.

After 4 week intervention period, metabolic response after feeding is significantly different between a follow-on formula containing low glycaemic carbohydrate and a conventional follow-on formula containing higher glycaemic carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy infants born
* weight between 10th and 90th percentile for age, according to the EURO Growth guidelines
* age between 5 - 7th month of life at study entry
* fully formula fed for at least 4 weeks before intervention start
* parents/caregivers understand the German language and are able to fill out questionnaires
* parents/caregivers agree to study participation and sign the informed consent form

Exclusion Criteria:

* acute or chronic illness of infant or mother
* drug and/or alcohol abuses of mother
* chronic medication
* participation of the infant in another intervention study
* gestational diabetes of the mother

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
metabolic response | After 4 week intervention period
  After 4 week intervention period, metabolic response after feeding is significantly different between a follow-on formula containing low glycaemic carbohydrate and a conventional follow-on formula containing higher glycaemic carbohydrates.

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Study Director — Germany, Hauner Childrens Hospital, Ludwig-Maximilians - University of Munich; Berthold Koletzko, Prof., Principal Investigator — Germany, Hauner Childrens Hospital, Ludwig-Maximilians - University of Munich
Locations (1):
- Germany, Hauner Childrens Hospital, Ludwig-Maximilians - University of Munich, Munich, Germany

REFERENCES:
- [Derived] Fleddermann M, Rauh-Pfeiffer A, Demmelmair H, Holdt L, Teupser D, Koletzko B. Effects of a Follow-On Formula Containing Isomaltulose (Palatinose) on Metabolic Response, Acceptance, Tolerance and Safety in Infants: A Randomized-Controlled Trial. PLoS One. 2016 Mar 17;11(3):e0151614. doi: 10.1371/journal.pone.0151614. eCollection 2016. PMID 26987056